CLINICAL TRIAL: NCT04334772
Title: Effectiveness of Percutaneous Microelectrolysis and Stretching Exercises on Agility, Strength, and Knee Joint Range in Hamstring Tightness in Athletes
Brief Title: Percutaneous Microelectrolysis in Agility, Joint Range and Strength
Acronym: MEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 603042020
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Hamstring Contractures
Keywords: Electric Stimulation Therapy; Electrolysis; Muscle Stretching Exercises; Muscle Strength; Agility; Hamstring Muscles
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle belly Microelectrolysis (Experimental): Group to receive direct current application percutaneously using an acupuncture needle with intensities in microamps (µA) at hamstring muscular belly. The acupuncture needle will correspond to the negative electrode or cathode.
  The group will also receive a passive stretching exercise treatment by a physical therapist.
  Interventions: Device: Muscle belly Microelectrolysis; Other: Stretching exercises
- Tendon Microelectrolysis (Experimental): Group to receive direct current application percutaneously using an acupuncture needle with intensities in microamps (µA) at the hamstring tendon. The acupuncture needle will correspond to the negative electrode or cathode.
  The group will also receive a passive stretching exercise treatment by a physical therapist.
  Interventions: Device: Tendon Microelectrolysis; Other: Stretching exercises
- Control (Active Comparator): Group to receive treatment by assisted passive stretching performed by a physical therapist on tightness hamstrings.
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Device: Muscle belly Microelectrolysis — three applications of direct current at 600 µA interrupted by intervals of 30 seconds between application at the level of the muscular belly of the shortened hamstrings.
  Arms: Muscle belly Microelectrolysis
Device: Tendon Microelectrolysis — three applications of direct current at 600 µA interrupted by intervals of 30 seconds between application in the tendon of the shortened hamstrings.
  Arms: Tendon Microelectrolysis
Other: Stretching exercises — 5 sets of passive static hamstring stretches using the straight leg extension (SLR) test for a time of 30 seconds and interval of 30 seconds for each

SUMMARY:
Electrical stimulation has a wide range of clinical applications in rehabilitation, being used for activities such as strengthening, pain control, management of edema, or control of inflammation after injury or surgery. One of the most classic forms of electrotherapy is direct current (DC), which stands out for its particular effects and which are not achieved with other forms of electrical stimulation.

A new therapeutic alternative through DC is Percutaneous Microelectrolysis (MEP), which began to have a significant boom in Latin America a couple of years ago. MEP is a minimally invasive procedure in which a low intensity DC is used. MEP has been proposed as a therapeutic resource to reduce muscle contractions and shortenings, thus favoring flexibility, although research to support this effect is lacking.

Muscle flexibility is an important component in rehabilitation and training programs. In lower limbs, tightness hamstring muscles is a common condition that limits flexibility and affects sedentary and athletic people. Loss of flexibility of hamstrings has been reported for different sports disciplines, showing a decrease in a high percentage with the exception of sports such as rhythmic gymnastics and dance where flexibility is essential for good performance. Loss of hamstring extensibility has been associated with a higher incidence of muscle tears, patellar tendinopathy, low back pain and alterations in lumbopelvic rhythm associated with compensatory biomechanical changes such as limb shortening, pelvic retroversion, and increased thoracic kyphosis, among others.

It is interesting to investigate the effectiveness of MEP in hamstring tightness. A increase in hamstring flexibility can contribute to increased joint range, muscle strength, and lower limb agility.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Electrotherapy is a valuable therapeutic resource used by physiotherapists for different purposes, among which are the reduction of pain, control of edema, muscle strengthening, control of the inflammatory process and promotion of tissue repair processes.[1,2] Within the The most widely used electrotherapy modalities are Sensory Transcutaneous Electrical Stimulation (TENS) and Burst Modulated Medium Frequency Alternating Currents (BMAC) commonly applied for analgesic purposes or for neuromuscular electrical stimulation (NMES).[2,3,4] Electromedicine also offers a variety of unidirectional currents such as direct (DC) or galvanic current and other low-frequency variants with a galvanic component such as diadynamic currents, 2-5 (Träbert), or faradic applications. [2,5 ] Direct current, described by Alexander Volta at the end of the 18th century, constitutes one of the first therapeutic currents, and has gained popularity in the last decade due to its use in percutaneous electrical applications that seek to promote tissue repair and decrease pain in musculoskeletal conditions. [5-10] DC is characterized by a unidirectional charge flow, of low voltage (60 to 80 volts) and constant intensity, and is produced from batteries or the rectification of alternating current from the electrical network. DC has particular physiological effects that are not achieved with other types of currents due to their physical characteristics. Its effects are based on the electrolysis process, a chemical decomposition phenomenon of some substances in solution subjected to a direct current and which results in electrophoresis (ion migration) and the formation of acidic or basic substances. [1,11-14] DC favors the accumulation of ions and charged molecules in the biological tissues that underlie the electrodes where it is applied. The deposition of charges occurs as a result of the electric forces of attraction and repulsion that are triggered by molecular dissociation, ionic migration, and accumulation of positive or negative charge depending on the electrode. All unidirectional currents are capable of greater or Less measure of producing electrophoresis and electrolysis under its poles (anode and cathode), triggering a series of physiological effects under the electrodes known as polar effects. These effects occur due to the modification of the local tissue pH and are directly related to the intensity of the current (mA) and its application time (minutes). Acidification of the medium by the production of substances such as hydrochloric acid (HCl) or carbonic acid (H2CO3), in addition to arteriolar vasoconstriction, hyperpolarization of neurons and coagulation, while alkalinization, caustic reactions due to the production of sodium hydroxide (NaOH), vasodilation, facilitation, depolarization and blood liquefaction occur at the cathode. [5,11-15] Due to its electrolytic effects, DC can cause chemical burns if its dosage is inadequate. This is how DC applications use intensities of the order of 0.05 µA/cm2 at 1mA/cm2, and treatment times between 12 to 15 minutes, although for iontophoresis applications, application of drugs loaded with tr Ascutaneous by means of DC, times of up to 30 or 40 minutes can be reached, although with maximum current intensities between 2 to 4mA. This dosage follows the recommendations of the literature to avoid potential adverse effects such as acid or alkaline burns. [5,12,15,19] The stratum corneum of human skin, on the other hand, constitutes an important barrier for bidirectional electric currents, offering a high impedance. although this response is dependent on intensity and time. It is the changes in skin impedance that ensure a depth of 4 to 5 cm for CD, a phenomenon that supports iontophoresis applications or electroporation treatments for drug delivery.[16,20,21]

   Percutaneous Microelectrolysis (MEP) In the last decade, different percutaneous procedures have emerged through DC that seek to induce electrolysis in deep musculoskeletal tissues.[6-9,24-26] An example of these percutaneous modalities is percutaneous microelectrolysis (MEP), which consists of the application of a microgalvanic current through acupuncture needles and where high current densities are achieved in the tissues due to the smaller surface area of the needle (2.5 to 3.8 mA/cm2). Unlike other electrolysis treatments, MEP has reported less discomfort in patients because microgalvanic currents (intensities less than 1 mA) are used in it. MEP uses the acupuncture needle (active electrode) as a cathode to induce in the tissues the synthesis of caustic substances such as sodium hydroxide (NaOH) or potassium hydroxide (KOH) resulting from the interaction of sodium (Na+2) and potassium (K+) ions with water (H2O) molecules. This promotes a controlled acute inflammatory response coupled with the release of molecular hydrogen or dihydrogen (H2) that inhibits free radicals that are concentrated in damaged musculoskeletal tissues. The analgesic effects of MEP are explained by the destruction of local free nerve endings as a consequence of the caustic response of the cathode. On the other hand, the needle's own mechanical stimulation promotes tissue micro-rupture that enhances the proinflammatory physiological effects of galvanism. Controlled inflammation induced by MEP promotes collagen genesis and increased circulation, initiating a new repair process Tissue. MEP is currently used as a treatment for acute and chronic tendon injuries, muscle injuries, and in the dermatofunctional area for the management of wrinkles, stretch marks, fibrosis and neuropathic scars. MEP has been proposed as a resource Therapeutic to reduce muscle contractions and shortenings, thus favoring flexibility, although there is a lack of research to support this effect.[24-30]

   Muscle flexibility Muscle flexibility is an important component in rehabilitation and training programs. In the lower limb, hamstring muscle shortening is a recurrent condition, a common condition that limits flexibility and affects sedentary, physically active, and athletic people. Hamstring flexibility is frequently evaluated in clinical tests and sports training, and is considered a component Basic physical abilities. Loss of flexibility of the hamstrings is associated with short-run sports and those in which knee flexion is favored, such as skiing, soccer, rugby, basketball, tennis, judo and volleyball.[31,32,33] Loss of hamstring flexibility has been reported for different sports disciplines, showing a decrease in a high percentage except for sports such as rhythmic gymnastics and dance where flexibility is essential for good performance.

   Hamstring tightness is characterized by a length-tension alteration compromising the articular range of hip flexion and knee extension, also associated with imbalances of muscular strength of the quadriceps-hamstring complex, which has been reported in soccer players. [31-35] Loss hamstring extensibility has been associated with a higher incidence of muscle tears, patellar tendinopathy, low back pain, and alterations in the lumbar-pelvic rhythm associated with compensatory biomechanical changes such as limb shortening, pelvic retroversion, and increased thoracic kyphosis. In addition, studies in soccer players have documented that a limitation in hamstring flexibility can compromise vertical jump, kick speed, short stroke and agility.

   Among the clinical tests used to evaluate hamstring tightness, the tests of straight leg elevation (Straight Leg Raising or SLR) and active knee extension (Active Knee Extension or AKE) stand out, the former demonstrating an intraclass reliability of 0.94 and the second an inter-examiner reliability of 0.99 (r). SLR is also used as a neurodynamic maneuver and as a test for clinical diagnosis of lumbar radiculopathy, lumbar hernia or sciatica, demonstrating a sensitivity of 0.67 and a specificity of 0.26. [31,34,40,41] Loss of hamstring extensibility is considered a modifiable risk variable and can be treated to prevent muscle injuries, especially if hamstring tear is considered to be one of the most frequent injuries in the athlete population and physically active people. In this sense, physical therapy has different intervention strategies to recover or improve flexibility, highlighting stretching exercises, soft tissue mobilization techniques, muscle energy techniques (PNF), neurodynamic sliding, electrical muscle elongation, dry puncture or thermotherapy modalities, although most of them have a short-lasting effect if they are not maintained over time. However, the static stretching strategy is the most used by physical therapists, sports trainers and physical educators, demonstrated good results in short and long or term.[31,49,50-52]
2. OBJECTIVES

   2.1. General purpose

   To assess the effectiveness of the Percutaneous Microelectrolysis (MEP) technique and stretching exercises in increasing agility, hamstring and quadriceps strength, and knee extension range in athletes with hamstring tightness.

   2.2. Specific objectives.
   * To assess differences in agility, hamstring and quadriceps strength, and knee extension joint range in the group exposed to muscle microelectrolysis between sessions.
   * To assess differences in agility, hamstring and quadriceps strength, and knee extension joint range in the group exposed to tendon microelectrolysis between sessions.
   * Compare the differences in agility, hamstring and quadriceps strength, and knee extension joint range between the groups exposed to microelectrolysis and the group treated with a stretching exercise plan for the intervention sessions.

   2.3. Investigation hypothesis

   Groups undergoing Percutaneous Microelectrolysis (MEP) at the level of the muscular and tendon belly will exhibit greater agility, hamstring and quadriceps strength, and increased knee extension joint range compared to the group treated with a stretching exercise plan.

   2.4. Hypothesis
   * H0: There will be no difference in agility, hamstring and quadriceps strength, and increased knee extension joint range between the group operated on with Percutaneous Microelectrolysis (MEP) and the group treated with a stretching exercise plan.
   * H1: Groups operated on with Percutaneous Microelectrolysis (MEP) will exhibit greater agility, hamstring and quadriceps strength, and increased knee extension joint range compared to the group treated with a stretching exercise plan.
3. METHODOLOGICAL DESIGN

   3.1. Type of study

   Experimental study, randomized clinical trial (RCT). Participants will be divided through a simple randomization process into three study groups; group 1 (application of microelectrolysis in the muscular belly), group 2 (application of microelectrolysis at the tendon level in the hamstrings) and group 3 (control).

   3.2. Ethical considerations of research

   The study will be presented to the Ethics Committee of the Eastern Metropolitan Health Service (SSMO) following the protocol of the principles of the Declaration of Helsinki. An informed consent will be applied to the participants in which the protocol and all the procedures of intervention. It will be made explicit in writing and verbally that the confidentiality of the data will be kept absolute, that participation will be voluntary and that the participants are free to leave the study at any time.

   3.3. Variables

   3.3.1 Conceptual definition of the variables.
   * Agility: Precise acceleration and deceleration movements and direction changes in the shortest possible time in seconds (sec) for the Agility T-Test. The test will consist of two attempts recording the shortest of the times obtained as the final value.
   * Muscular strength: Maximum isometric strength (FIMáx) of shortened hamstrings and ipsilateral femoral quadriceps developed over 4 to 6 seconds, obtained from the best of three attempts in a voluntary maximum contraction. Hamstring and quadriceps strength will be assessed with electromechanical dynamometry on a quadriceps table with the participant seated keeping his knee flexed 90° and anchoring the dynamometer pulley at the distal end of the leg.
   * Knee joint range: Maximum active range of knee extension performed with the limb shortened in the supine position from a 90° hip flexion and 90° knee flexion.
   * Percutaneous microelectrolysis (MEP): Direct current application percutaneously using an acupuncture needle with intensities in microamps (µA) at the level of the muscular belly or hamstring tendon. The acupuncture needle will correspond to the negative electrode or cathode.
   * Stretching exercise: Passive assisted stretching performed by a physical therapist on the shortened hamstrings. The stretch will be performed with the participant in the supine position through the straight leg extension test (SLR), perceiving the point of maximum hamstring tension and keeping the limb at that point for 30 seconds.

   3.3.2. Operational definition of variables.
   * Agility: Agility will be quantified as the minimum time in seconds (sec) that the participant takes to complete the circuit for the Agility T-Test.
   * Muscular strength: The strength of the hamstrings and femoral quads will be evaluated with the Dynasystem functional electromechanical dynamometer (DEMF) from the company Symotech (Madrid, Spain). The maximum isometric force shall be recorded in newtons (N).
   * Knee joint range: The active range of knee extension will be evaluated in degrees of extension using the Active Knee Extension Test (AKE) with a manual goniometer (APPENDIX 7). The lateral condyle of the femur will be taken as a fixed point, the fixed arm will remain parallel to the axis of the thigh and the mobile arm will project to the ipsilateral lateral malleolus.
   * Percutaneous microelectrolysis (MEP): CD will be applied with the SVELTIA® electro stimulator. The current dose (mA * min) applied to each participant will be recorded based on the current intensity (mA) and total therapeutic time (minutes). The protocol will include three 600 µA direct current applications interrupted by 30 second intervals between applications.
   * Stretching exercise: 5 sets of passive static hamstring stretches will be performed using the straight leg extension test (SLR) for a time of 30 seconds and an interval of 30 seconds for each series.

   3.3.3. Variable type definition.
   * Agility: Dependent, quantitative, ratio variable.
   * Muscular strength: Dependent, quantitative, ratio variable.
   * Knee joint range: Dependent, quantitative, interval variable.
   * Percutaneous microelectrolysis (MEP): Independent, quantitative, interval variable.
   * Stretching exercise: Independent variable, quantitative, ratio variable.
4. MATERIALS AND METHOD

   4.1. Participants

   For the study, the athletes from the Andrés Bello University belonging to the rugby, soccer, basketball or tennis teams will be considered as participants. An invitation will be made to all athletes through the institution's National Director of Sports, making it clear that participation is completely voluntary. Those interested will be contacted via email or telephone and will be summoned in person to explain the characteristics and objectives of the study. Subsequently, they will be asked to sign a consent, making explicit the voluntary participation and the withdrawal to continue at the time they determine.

   4.2 Aletorization and sample size.

   The participants will be evaluated according to the selection criteria (inclusion and exclusion) through a survey with closed questions and a clinical examination in which the presence or absence of hamstring shortening will be determined, as well as its laterality. . Participants will be divided through a simple randomization process (table of random numbers) into three study groups; group 1 (application of microelectrolysis in the muscular belly), group 2 (application of microelectrolysis at the tendon level in the hamstrings) and group 3 (control). All groups will be called twice a week to carry out the assigned treatment. All groups will receive as a basic treatment a therapeutic exercise plan for static hamstring stretching of 5 series for 30 seconds twice a week, and groups 1 and 2 will receive in addition to the exercise plan an intervention of differentiated microelectrolysis (in the muscle belly or tendon).

   The sample size was determined from the effect size obtained by evidence reported for static stretching. Therefore the sample size is calculated as 10 subjects per group.

   4.3. Process

   Joint range of knee extension, maximum isometric muscle strength of quadriceps and hamstrings, and agility will be evaluated in all groups once a week. The study will last 4 weeks, so all groups will complete a total of 8 treatment sessions and 4 evaluation sessions. Joint range differences (ΔROM), maximum isometric muscle strength difference (ΔFImax) and agility difference (ΔAg) between the 4 sessions will be considered as main variables.

   4.4. Phases of the study

   Three phases have been designated for the investigation; 1. Sampling phase, 2. Evaluation phase and 3. Intervention phase. The sampling phase will consist of applying the selection survey to all athletes interested in participating in the study. The survey will be applied to those selected for rugby, soccer, basketball and tennis at Andrés Bello University through the Google Drive® system. All those who meet the survey selection criteria will be invited to participate in the research. This stage will last two weeks.

   The evaluation phase will last two weeks and will determine a second filter of the population. The athletes selected by the survey and who gave their written consent will participate in it. At this stage, a clinical examination will be performed to determine the presence of hypermobility using the Beighton hypermobility test and the presence of hamstring shortening through the Straight Leg Raising (SLR) test. An examiner will assess the presence of hypermobility in athletes to later assess the presence or absence of hamstring shortening. In relation to the Beighton test, a score greater than 5 will indicate the presence of hypermobility and will exclude the study participant. The SLR test will be performed using an inclinometer and will be considered a positive test when the participant reports tightness or tension in the back of the thigh when raising the limb with an angle less than 80° of hip flexion.If Both extremities have an elevation of less than 80°. The one with the lowest value will be considered short. Participants with a negative physical examination (-), that is, without the presence of hamstring shortening according to the protocol, will be excluded, while those with a positive physical examination (+) will become the definitive sample. The evaluator will record the laterality of the limb with the shortening in a Microsoft Excel® spreadsheet.

   The intervention phase will take place over a period of 10 weeks. The sample will be randomized into three working groups; group 1 (application of microelectrolysis in the muscular belly), group 2 (application of microelectrolysis at the tendon level in the hamstrings) and group 3 (control). The randomization of the sample will be performed by the study director using the simple random sampling process through a table of random numbers taken from the tables proposed by the RAND Corporation®. The study director will be the only one with access to the randomization table. Demographic variables (secondary variables) for each group, including age, sex and body mass index (BMI) will be tabulated in a Microsoft Excel® program spreadsheet.

   Participants in each group will be evaluated by three evaluators to determine knee extension basal joint range (ROMEXT), maximum isometric muscle strength for hamstrings and ipsilateral femoral quadriceps (FIImax and FICmax), and agility in (Ag). The range will be measured through goniometry, muscle strength will be evaluated by electromechanical dynamometry and agility will be determined through the T agility test.

   ROMEXT, FImax and Ag values will be evaluated in degrees (°), Newtons (N) and seconds (sec) respectively, and will be considered as primary variables of the study. ROMEXT, FImax and Ag will be tabulated in an Excel® spreadsheet for each evaluator. The evaluations will last 4 weeks, with one evaluation per week. Said evaluation will be carried out before and after the intervention assigned to each group. Participants will be called twice a week to carry out their corresponding treatments, making one of these visits coincide with the corresponding evaluation session for the current week.

   4.5. Statistical analysis

   The descriptive statistics for the primary variables ROMEXT, FImax and Ag will use as analysis measures, means and standard deviation (x, DS), or median and interquartile range (med, RIC). For secondary variables such as sex, body mass index (BMI), frequencies and averages or medians, respectively, will be used.

   Regarding inferential statistics, the SHAPIRO WILK (S-WILK) normality test will be used to determine if the distribution of data obtained for the primary and secondary variables is normal or not, and according to this, the statistical test atingente, test ANOVA if the data distributes normally or Kruskal Wallis test if the data does not distribute normal. The SPSS v.24.0 program will be used for the statistical calculation. Once the analysis is done, a month will be considered for the analysis of the results obtained, discussion approach and conclusion.
5. EVALUATION PROTOCOLS

5.1. Hypermobility Assessment - Beighton Hypermobility Test.

The Beighton test is a clinical test for the detection of ligament hypermobility or excessive joint range (joint hypermobility). The test requires having a score equal to 5 or higher of a total of 9 to be considered positive (+). Participants are evaluated on a 9-point scale, considering 1 point for each hypermobile site, performed bilaterally. The test includes the following points;

* Hyperextension of the elbows (greater than 10°), with the subject sitting on a stool and with the arm explored by the extension examiner (bilateral evaluation, 2 points).
* Passively touch the forearm with the thumb, holding the wrist in flexion, with the individual in the same position as the previous point (bilateral evaluation, 2 points).
* Passive extension of the index finger to more than 90°, with the participant sitting and with the palm of the hand fully resting on the table (bilateral evaluation, 2 points).
* Hyperextension of the knees (more than 100°), with the participant in supine position (bilateral evaluation, 2 points).
* Forward trunk flexion touching the ground with the palms of the hands when bending over without bending the knees (1 point).

Participants who give a positive Beighton test (+) will be excluded from the study this because joint hypermobility can generate false negative short hamstrings for evaluation.

5.2. Hamstring Shortening Assessment - Straight Leg Hip Flexion Test (SLR).

The evaluation will be performed using the straight leg hip flexion test (SLR). The straight leg lift is a passive test testing each limb individually. The participant will lie supine without a pillow under his head, while the examiner will stand on the side of the table. The evaluator will take the ankle and passively flex one of the hips keeping the knee in extension while the point of tension is perceived, accompanied by a sensation of tightness reported by the user. The angle formed between the surface of the stretcher and the axis of the lower limb will be measured. It will be considered as a positive test (+) if the degree of tension referred to with the test is less than 80°, while if the tension appears above 80° the negative test (-) will be considered. The test is compared with the contralateral side to determine the predominance of hamstring shortening. Possible findings when performing the test may include;

1. Neither limb has short hamstrings; SLR negative (-) bilaterally. The participant will be excluded by not completing the selection criteria.
2. One of the extremities has short hamstrings; Positive SLR (+) for one of the two extremities. The participant will be included in the research.
3. Both limbs drop short hamstrings; SLR positive bilaterally. The participant will be included in the research and the limb with the least degrees of elevation will be considered as the side with short hamstrings.

5.3. Joint Knee Range Assessment - Active Knee Extension Test (AKE).

The Active Knee Extension Test (AKE) is used to assess the length of the hamstrings and the range of active knee extension in the 90 ° hip flexion position. The participant will be placed in a supine position on a stretcher while maintaining one hip in 90° flexion and the knee in 90 ° flexion while the contralateral lower extremity is fully supported. The participant is instructed to perform an active maximum knee extension. The evaluator will measure the angle of extension from the knee flexion position of 90°, which will be considered as the 0 ° articular position from which the measurement will be recorded. The degrees of knee extension will be recorded using a manual goniometer.

5.4. Evaluation of muscular strength of hamstrings and femoral quadriceps.

Maximum voluntary isometric contraction of the knee flexor and extensor muscles will be assessed. Strength will be assessed through a functional electromechanical dynamometer (DEMF) on the side that was recorded with short hamstrings. For the evaluation, the participant will be placed on a quadriceps table keeping the knee in 90° flexion while fixing the thigh in its anterior distal part with a belt to avoid lifting the thigh during the test. The participant must keep his back supported during the test. For the record, the pulley will be anchored to the distal end of the leg, maintaining a 90° angle between the pulley and the leg. To record the hamstring strength, the pulley will be placed in front of the leg so that the participant flexes the knee and the rope perceives the degree of tension generated. To record the quadriceps force, the pulley will be anchored behind the leg so that when performing the knee extension the rope perceives the tension generated. Before the test, each subject will perform an adequate warm-up, consisting of 2 to 3 submaximal contractions to become familiar with the test procedure. Each subject will perform a maximum voluntary isometric contraction for hamstrings and femoral quads for 4 to 6 seconds in three series. 1 minute rest between attempts will be considered to avoid the effects of fatigue. During the test the subject will be instructed to exert as much force as possible.

5.5. Agility assessment - T Agility test (T Agility test).

The Agility T-Test is reliable and valid to measure the ability to quickly change directions and speed based on stops and agility. The test consists of various multidirectional displacements, running forward, laterally to the right and left. For the test, 4 cones (a, b, c and d) are used simulating the letter t. Three of them are placed at a lateral distance of 5 meters and another is placed 10 meters from the central cone. The participant will be instructed to run as fast as possible from the first cone (cone a) forward (cone b), then move laterally to the right (cone c), then laterally to the left (cone d), to return laterally to the cone b and run to the starting cone (cone a). Agility will be quantified as the minimum time in seconds (sec) that the participant takes to complete the circuit for the test. The test will be carried out in two attempts taking, registering the least of the times as the final value. A 2-minute break will be considered between attempts to avoid the effects of fatigue.

Before performing the agility test, a five-minute pre-heating will be carried out on a cycle ergometer (MONARK 915E®) at a power of 80 watts.

6. TREATMENT PROTOCOLS

6.1. Application of electrotherapy Percutaneous Microelectrolysis (MEP)

For the application of microelectrolysis, the SVELTIA® Direct Current equipment will be used. Acupuncture needles 0.3 millimeters thick and 25 millimeters long will be used.

The procedure will be performed with latex gloves to avoid any contact with the skin. The acupuncture needle will be inserted into the point of the muscular belly or hamstring tendon. It will work with an intensity of 0.6 milliamps (mA). It will be entered perpendicularly with the acupuncture needle mounted on the device's pointer with an emission of 100 microamps (µA). When it has been entered, the intensity will be increased to 600 µA and the participant will be told that when burning, pain or oppression appears, and that these discomforts become uncomfortable, notify the provider. The time of emission until the appearance of symptoms will be designated as T1. At that time the broadcast will be paused for 30 seconds. A second emission will be carried out maintaining the 600 µA until the participant again manifests a burning sensation or discomfort. The current application time will be recorded as T2. The 30 second pause will repeat. The third emission or T3 will be performed at the same time as the emission registered for T2 or until the person reports discomfort by withdrawing the needle to later finish the procedure.

After MEP, a reevaluation of the knee extension range (AKE test), hamstring and femoral quadriceps (functional electromechanical dynamometry) and agility test (T-Test) will be performed.

6.2 Passive static stretching application (group 1, 2 and 3).

The three groups will receive as a base treatment a hamstring stretching protocol for the limb evaluated with shortening. The stretch will be performed using the straight leg hip flexion test (SLR). The handler will raise the shortened lower limb to the point of maximum tension reported by the participant to keep it in that position. The stretches will consist of 5 sets of 30 seconds with a break between sets of 30 seconds, thus completing a 1-minute work cycle (stretching and resting). The time will begin to count after locating the stress angle.

After the intervention with stretching exercises for group 3 (control group), a reevaluation of the knee extension range (AKE test), hamstring and femoral quadriceps (functional electromechanical dynamometry) and agility test (T-Test) will be performed). On the other hand, once the stretching exercises for group 1 and 2 (muscular and tendon microelectrolysis) have been completed, a reevaluation of the knee extension range (AKE test), hamstring muscle strength and femoral quadriceps (functional electromechanical dynamometry) and agility test will be performed. (T-Test).

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years of age.
* Athletes from the university teams in the branches of rugby, soccer, basketball or tennis.
* Presence of hamstring shortening in one of the two extremities (positive straight leg elevation test or Straight Leg Raising). It will be considered as a positive test when the participant, in the supine position, shows tension or discomfort in the posterior region of the thigh when passively raising the lower limb for any angle less than 80 ° of hip flexion with extended knee. In the event that the participant presents a bilateral shortening, the limb with the lower elevation will be taken as shortened hamstrings.

Exclusion criteria.

* Pain when performing hip or knee movements.
* Musculoskeletal injuries such as fractures, sprains, tears, dislocations, contusions, or joint problems of the lower extremities in the past 3 months.
* Skin disorders such as scars, burns, psoriasis or wounds in the posterior region of the thighs.
* Neurological signs or symptoms such as tingling, loss of sensation in the lower extremities (partial or complete), weakness, changes in color or temperature in the thigh, legs or foot.
* Background or circulatory abnormalities in the lower extremities such as arterial ischemia, venous insufficiency, embolism, post-phlebitic syndrome, lymphedema or deep vein thrombosis.
* Joint hypermobility (positive Beighton hypermobility test).
* Intake of medications or anti-inflammatory drug treatment at the time of recruitment (includes non-steroidal or steroidal anti-inflammatory drugs).
* Allergy to metals.
* Apprehension or fear of the application of electric current.
* Belonephobia (extreme and uncontrollable fear of needles and other objects that can cause bloody wounds such as pins, knives, pocket knives, syringes, etc.).

Elimination criteria.

* Discomfort during the intervention with electrotherapy that requires stopping treatment.
* Failure to complete the evaluation protocol (attendance at all scheduled evaluation sessions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Maximum isometric strength differences | Baseline and 2 hours later (1 session of treatment)
  Comparing maximum hamstring isometric strength changes pre and post application of microelectrolysis and hamstring stretching protocol.
Joint Range differences | Baseline and 2 hours later (1 session of treatment)
  Comparing maximum knee extention range pre and post application of microelectrolysis and hamstring stretching protocol.
Agility differences | Baseline and 2 hours later (1 session of treatment)
  Comparison of time changes in performing the T agility test pre and post application of microelectrolysis and hamstring stretching protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hernán A de la Barra, Msc, Principal Investigator — Universidad Andrés Bello
Locations (1):
- Universidad Andrés Bello, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadil V, Sadil S. [Electrotherapy]. Wien Med Wochenschr. 1994;144(20-21):509-20. German. PMID 7879402
- [Background] Samuel SR, Maiya GA. Application of low frequency and medium frequency currents in the management of acute and chronic pain-a narrative review. Indian J Palliat Care. 2015 Jan-Apr;21(1):116-20. doi: 10.4103/0973-1075.150203. PMID 25709199
- [Background] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- [Background] Lopez-Martos R, Gonzalez-Perez LM, Ruiz-Canela-Mendez P, Urresti-Lopez FJ, Gutierrez-Perez JL, Infante-Cossio P. Randomized, double-blind study comparing percutaneous electrolysis and dry needling for the management of temporomandibular myofascial pain. Med Oral Patol Oral Cir Bucal. 2018 Jul 1;23(4):e454-e462. doi: 10.4317/medoral.22488. PMID 29924769
- [Background] Fernandez-Rodriguez T, Fernandez-Rolle A, Truyols-Dominguez S, Benitez-Martinez JC, Casana-Granell J. Prospective Randomized Trial of Electrolysis for Chronic Plantar Heel Pain. Foot Ankle Int. 2018 Sep;39(9):1039-1046. doi: 10.1177/1071100718773998. Epub 2018 May 17. PMID 29771148
- [Background] Mattiussi G, Moreno C. Treatment of proximal hamstring tendinopathy-related sciatic nerve entrapment: presentation of an ultrasound-guided "Intratissue Percutaneous Electrolysis" application. Muscles Ligaments Tendons J. 2016 Sep 17;6(2):248-252. doi: 10.11138/mltj/2016.6.2.248. eCollection 2016 Apr-Jun. PMID 27900300
- [Background] Abat F, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Clinical results after ultrasound-guided intratissue percutaneous electrolysis (EPI(R)) and eccentric exercise in the treatment of patellar tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1046-52. doi: 10.1007/s00167-014-2855-2. Epub 2014 Jan 30. PMID 24477495
- [Background] Rampazo da Silva EP, da Silva VR, Bernardes AS, Matuzawa FM, Liebano RE. Study protocol of hypoalgesic effects of low frequency and burst-modulated alternating currents on healthy individuals. Pain Manag. 2018 Mar;8(2):71-77. doi: 10.2217/pmt-2017-0058. Epub 2018 Feb 16. PMID 29451431
- [Background] Dolhem R. [The history of electrostimulation in rehabilitation medicine]. Ann Readapt Med Phys. 2008 Jul;51(6):427-31. doi: 10.1016/j.annrmp.2008.04.004. Epub 2008 May 21. French. PMID 18539356
- [Background] Piccolino M. Luigi Galvani's path to animal electricity. C R Biol. 2006 May-Jun;329(5-6):303-18. doi: 10.1016/j.crvi.2006.03.002. Epub 2006 Mar 30. PMID 16731488
- [Background] Piccolino M. Luigi Galvani and animal electricity: two centuries after the foundation of electrophysiology. Trends Neurosci. 1997 Oct;20(10):443-8. doi: 10.1016/s0166-2236(97)01101-6. PMID 9347609
- [Background] Kalia YN, Naik A, Garrison J, Guy RH. Iontophoretic drug delivery. Adv Drug Deliv Rev. 2004 Mar 27;56(5):619-58. doi: 10.1016/j.addr.2003.10.026. PMID 15019750
- [Background] Ita K. Transdermal iontophoretic drug delivery: advances and challenges. J Drug Target. 2016;24(5):386-91. doi: 10.3109/1061186X.2015.1090442. Epub 2015 Sep 25. PMID 26406291
- [Background] Conjeevaram R, Banga AK, Zhang L. Electrically modulated transdermal delivery of fentanyl. Pharm Res. 2002 Apr;19(4):440-4. doi: 10.1023/a:1015135426838. PMID 12033377
- [Background] Kalia YN, Guy RH. The electrical characteristics of human skin in vivo. Pharm Res. 1995 Nov;12(11):1605-13. doi: 10.1023/a:1016228730522. PMID 8592657
- [Background] Prausnitz MR, Langer R. Transdermal drug delivery. Nat Biotechnol. 2008 Nov;26(11):1261-8. doi: 10.1038/nbt.1504. PMID 18997767
- [Background] Ferreira ACR, Guida ACP, Piccini AA, Parisi JR, Sousa L. Galvano-puncture and dermabrasion for striae distensae: a randomized controlled trial. J Cosmet Laser Ther. 2019;21(1):39-43. doi: 10.1080/14764172.2018.1444777. Epub 2018 Mar 16. PMID 29547019
- [Background] Espejo-Antunez L, Lopez-Minarro PA, Garrido-Ardila EM, Castillo-Lozano R, Dominguez-Vera P, Maya-Martin J, Albornoz-Cabello M. A comparison of acute effects between Kinesio tape and electrical muscle elongation in hamstring extensibility. J Back Musculoskelet Rehabil. 2015;28(1):93-100. doi: 10.3233/BMR-140496. PMID 25061028
- [Background] Henderson G, Barnes CA, Portas MD. Factors associated with increased propensity for hamstring injury in English Premier League soccer players. J Sci Med Sport. 2010 Jul;13(4):397-402. doi: 10.1016/j.jsams.2009.08.003. Epub 2009 Oct 2. PMID 19800844
- [Background] Reid DA, McNair PJ. Passive force, angle, and stiffness changes after stretching of hamstring muscles. Med Sci Sports Exerc. 2004 Nov;36(11):1944-8. doi: 10.1249/01.mss.0000145462.36207.20. PMID 15514511
- [Background] Freckleton G, Pizzari T. Risk factors for hamstring muscle strain injury in sport: a systematic review and meta-analysis. Br J Sports Med. 2013 Apr;47(6):351-8. doi: 10.1136/bjsports-2011-090664. Epub 2012 Jul 4. No abstract available. PMID 22763118
- [Background] Mason JS, Crowell M, Dolbeer J, Morris J, Terry A, Koppenhaver S, Goss DL. THE EFFECTIVENESS OF DRY NEEDLING AND STRETCHING VS. STRETCHING ALONE ON HAMSTRING FLEXIBILITY IN PATIENTS WITH KNEE PAIN: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2016 Oct;11(5):672-683. PMID 27757280
- [Background] Kim DH, Lee JJ, Sung Hyun You J. Effects of instrument-assisted soft tissue mobilization technique on strength, knee joint passive stiffness, and pain threshold in hamstring shortness. J Back Musculoskelet Rehabil. 2018;31(6):1169-1176. doi: 10.3233/BMR-170854. PMID 30040707
- [Background] Fousekis K, Tsepis E, Poulmedis P, Athanasopoulos S, Vagenas G. Intrinsic risk factors of non-contact quadriceps and hamstring strains in soccer: a prospective study of 100 professional players. Br J Sports Med. 2011 Jul;45(9):709-14. doi: 10.1136/bjsm.2010.077560. Epub 2010 Nov 30. PMID 21119022
- [Background] Devan MR, Pescatello LS, Faghri P, Anderson J. A Prospective Study of Overuse Knee Injuries Among Female Athletes With Muscle Imbalances and Structural Abnormalities. J Athl Train. 2004 Sep;39(3):263-267. PMID 15496997
- [Background] Araki T, Kato H, Kogure K. Protective effect of vinconate, a novel vinca alkaloid derivative, on glucose utilization and brain edema in a new rat model of middle cerebral artery occlusion. Gen Pharmacol. 1992 Jan;23(1):141-6. doi: 10.1016/0306-3623(92)90061-n. PMID 1592223
- [Background] Geist K, Bradley C, Hofman A, Koester R, Roche F, Shields A, Frierson E, Rossi A, Johanson M. Clinical Effects of Dry Needling Among Asymptomatic Individuals With Hamstring Tightness: A Randomized Controlled Trial. J Sport Rehabil. 2017 Nov;26(6):507-517. doi: 10.1123/jsr.2016-0095. Epub 2016 Nov 11. PMID 27834590
- [Background] Hui SS, Yuen PY. Validity of the modified back-saver sit-and-reach test: a comparison with other protocols. Med Sci Sports Exerc. 2000 Sep;32(9):1655-9. doi: 10.1097/00005768-200009000-00021. PMID 10994920
- [Background] Garcia-Pinillos F, Ruiz-Ariza A, Moreno del Castillo R, Latorre-Roman PA. Impact of limited hamstring flexibility on vertical jump, kicking speed, sprint, and agility in young football players. J Sports Sci. 2015;33(12):1293-7. doi: 10.1080/02640414.2015.1022577. Epub 2015 Mar 12. PMID 25761523
- [Background] Neto T, Jacobsohn L, Carita AI, Oliveira R. Reliability of the Active-Knee-Extension and Straight-Leg-Raise Tests in Subjects With Flexibility Deficits. J Sport Rehabil. 2015 Dec 3;24(4):2014-0220. doi: 10.1123/jsr.2014-0220. Print 2015 Nov 1. PMID 25364856
- [Background] Cameron DM, Bohannon RW. Relationship between active knee extension and active straight leg raise test measurements. J Orthop Sports Phys Ther. 1993 May;17(5):257-60. doi: 10.2519/jospt.1993.17.5.257. PMID 8343784
- [Background] Rabin A, Gerszten PC, Karausky P, Bunker CH, Potter DM, Welch WC. The sensitivity of the seated straight-leg raise test compared with the supine straight-leg raise test in patients presenting with magnetic resonance imaging evidence of lumbar nerve root compression. Arch Phys Med Rehabil. 2007 Jul;88(7):840-3. doi: 10.1016/j.apmr.2007.04.016. PMID 17601462
- [Background] Deville WL, van der Windt DA, Dzaferagic A, Bezemer PD, Bouter LM. The test of Lasegue: systematic review of the accuracy in diagnosing herniated discs. Spine (Phila Pa 1976). 2000 May 1;25(9):1140-7. doi: 10.1097/00007632-200005010-00016. PMID 10788860
- [Background] Medeiros DM, Cini A, Sbruzzi G, Lima CS. Influence of static stretching on hamstring flexibility in healthy young adults: Systematic review and meta-analysis. Physiother Theory Pract. 2016 Aug;32(6):438-445. doi: 10.1080/09593985.2016.1204401. Epub 2016 Jul 26. PMID 27458757
- [Background] Hopper D, Deacon S, Das S, Jain A, Riddell D, Hall T, Briffa K. Dynamic soft tissue mobilisation increases hamstring flexibility in healthy male subjects. Br J Sports Med. 2005 Sep;39(9):594-8; discussion 598. doi: 10.1136/bjsm.2004.011981. PMID 16118294
- [Background] Shadmehr A, Hadian MR, Naiemi SS, Jalaie S. Hamstring flexibility in young women following passive stretch and muscle energy technique. J Back Musculoskelet Rehabil. 2009;22(3):143-8. doi: 10.3233/BMR-2009-0227. PMID 20023343
- [Background] Oranchuk DJ, Flattery MR, Robinson TL. Superficial heat administration and foam rolling increase hamstring flexibility acutely; with amplifying effects. Phys Ther Sport. 2019 Nov;40:213-217. doi: 10.1016/j.ptsp.2019.10.004. Epub 2019 Oct 7. PMID 31605900
- [Background] Decoster LC, Cleland J, Altieri C, Russell P. The effects of hamstring stretching on range of motion: a systematic literature review. J Orthop Sports Phys Ther. 2005 Jun;35(6):377-87. doi: 10.2519/jospt.2005.35.6.377. PMID 16001909
- [Background] Fakhro MA, Chahine H, Srour H, Hijazi K. Effect of deep transverse friction massage vs stretching on football players' performance. World J Orthop. 2020 Jan 18;11(1):47-56. doi: 10.5312/wjo.v11.i1.47. eCollection 2020 Jan 18. PMID 31966969
- [Background] Koklu Y, Alemdaroglu U, Kocak FU, Erol AE, Findikoglu G. Comparison of chosen physical fitness characteristics of Turkish professional basketball players by division and playing position. J Hum Kinet. 2011 Dec;30:99-106. doi: 10.2478/v10078-011-0077-y. Epub 2011 Dec 25. PMID 23486863
- [Background] Cini A, de Vasconcelos GS, Lima CS. Acute effect of different time periods of passive static stretching on the hamstring flexibility. J Back Musculoskelet Rehabil. 2017;30(2):241-246. doi: 10.3233/BMR-160740. PMID 27472859
- [Background] Fessi MS, Makni E, Jemni M, Elloumi M, Chamari K, Nabli MA, Padulo J, Moalla W. Reliability and criterion-related validity of a new repeated agility test. Biol Sport. 2016 Jun;33(2):159-64. doi: 10.5604/20831862.1198635. Epub 2016 Apr 2. PMID 27274109
- [Background] Freitas TT, Calleja-Gonzalez J, Alarcon F, Alcaraz PE. Acute Effects of Two Different Resistance Circuit Training Protocols on Performance and Perceived Exertion in Semiprofessional Basketball Players. J Strength Cond Res. 2016 Feb;30(2):407-14. doi: 10.1519/JSC.0000000000001123. PMID 26813631
- [Background] Rodriguez-Perea A, Chirosa Rios LJ, Martinez-Garcia D, Ulloa-Diaz D, Guede Rojas F, Jerez-Mayorga D, Chirosa Rios IJ. Reliability of isometric and isokinetic trunk flexor strength using a functional electromechanical dynamometer. PeerJ. 2019 Oct 18;7:e7883. doi: 10.7717/peerj.7883. eCollection 2019. PMID 31695965
- [Background] Jerez-Mayorga D, Chirosa Rios LJ, Reyes A, Delgado-Floody P, Machado Payer R, Guisado Requena IM. Muscle quality index and isometric strength in older adults with hip osteoarthritis. PeerJ. 2019 Aug 7;7:e7471. doi: 10.7717/peerj.7471. eCollection 2019. PMID 31410316
- [Background] Takahashi Y, Yamaji T. Comparison of effects of joint flexibility on the lumbo-pelvic rhythm in healthy university students while bending the trunk forward. J Phys Ther Sci. 2020 Mar;32(3):233-237. doi: 10.1589/jpts.32.233. Epub 2020 Mar 11. PMID 32184539
- [Background] Ong JH, Lim J, Chong E, Tan F. The Effects of Eccentric Conditioning Stimuli on Subsequent Counter-Movement Jump Performance. J Strength Cond Res. 2016 Mar;30(3):747-54. doi: 10.1519/JSC.0000000000001154. PMID 26332775
- [Background] Alizadeh Ebadi L, Cetin E. Duration Dependent Effect of Static Stretching on Quadriceps and Hamstring Muscle Force. Sports (Basel). 2018 Mar 13;6(1):24. doi: 10.3390/sports6010024. PMID 29910328